CLINICAL TRIAL: NCT04283656
Title: A Prospective, Randomized, Three-period Crossover, Interaction Study to Evaluate the Pharmacokinetics of Doravirine and Tenofovir Disoproxil Fumarate Co-administered With Cross-sex Hormonal Therapy in Adult HIV-negative Transgender Women
Brief Title: Evaluating Drug Interactions Between Doravirine With Estradiol and Spironolactone in Healthy Transgender Women
Acronym: IDENTIFY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Walter K. Kraft, Principal Investigator, Thomas Jefferson University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15431
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Transgender Health; Gender Dysphoria; Transgender Women; Human Immunodeficiency Virus
MeSH Terms: conditions — Gender Dysphoria; Acquired Immunodeficiency Syndrome | interventions — doravirine; Canrenoic Acid; Spironolactone; Estradiol

STUDY DESIGN:
Intervention Model Description: Three period crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment A (Experimental): Single-dose oral Doravirine/lamivudine/tenofovir disoproxil
  Interventions: Drug: Doravirine/Lamivudine/Tenofovir
- Treatment B (Experimental): Single-dose estradiol and spironolactone co-administered with placebo
  Interventions: Drug: Spironolactone 100mg; Drug: Estradiol 2mg; Other: Placebo
- Treatment C (Experimental): Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone
  Interventions: Drug: Doravirine/Lamivudine/Tenofovir; Drug: Spironolactone 100mg; Drug: Estradiol 2mg

INTERVENTIONS:
Drug: Doravirine/Lamivudine/Tenofovir — 100mg/300mg/300mg orally for one dose, daily
  Other Names: Delstrigo
  Arms: Treatment A; Treatment C
Drug: Spironolactone 100mg — 200mg orally for two doses, twice-daily
  Other Names: Aldactone
  Arms: Treatment B; Treatment C
Drug: Estradiol 2mg — 4mg orally for two doses, twice-daily
  Arms: Treatment B; Treatment C
Other: Placebo — Placebo for one dose, daily
  Arms: Treatment B

SUMMARY:
Transgender women living with Human Immunodeficiency Virus (HIV) may prioritize gender-affirming hormonal therapy over antiretroviral drug therapy. Hormonal therapy typically consists of oral estradiol and spironolactone, which induce drug-metabolizing enzymes after prolonged administration. This study evaluates the bi-directional potential drug interaction between the antiretroviral drug, doravirine, when co-administered with estradiol and spironolactone.

DETAILED DESCRIPTION:
This study will consist of healthy transgender women volunteers randomized to a 1:1 sequence ("E" or "F") There are three periods and in each period there are one of three treatments

Treatment A: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate alone Treatment B: Single-dose estradiol and spironolactone co-administered with placebo Treatment C: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone

The primary outcome measures are the drug concentrations

The primary comparisons are geometric mean ratios of drugs with potential perpetrators of drug interactions using a crossover method

ELIGIBILITY:
Inclusion Criteria:

* Healthy self-identified transgender women (male-to-female) between 18-45 years old at the time of screening
* Have not undergone an orchiectomy
* Receiving oral estradiol and spironolactone for >/= 3 months prior to study entry with a self-reported adherence to prescribed doses of >/= 90%
* Agree to abstain from alcohol consumption throughout the duration of the study
* Be willing to briefly interrupt hormonal therapy prior to and during the study
* If on pre-exposure prophylaxis (PrEP) therapy containing tenofovir alafenamide or tenofovir disoproxil fumarate, willing to discontinue PrEP at least 2 weeks before study start and for the duration of the study
* Agree to use condoms for all sexual activity prior to the start and throughout the duration of the study
* Evidence of a personal signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Presence of clinically significant acute or chronic disease, that in the investigator's opinion, would compromise the participant's safety during the study
* Use of injectable or transdermal estradiol
* Use of any other hormonal replacement therapy, wit h the exception of oral estradiol and spironolactone
* Current use of any antiretroviral drug. This will not be exclusionary if participants reported discontinuing within 30 days of screening
* Creatinine clearance </= 60 mL/min, as estimated by the Cockcroft-Gault equation
* Known anaphylactic or severe systemic reactions to any components of doravirine, lamivudine, or tenofovir disoproxil fumarate
* Positive HIV, hepatitis B or Hepatitis C virus at screening. Evidence of prior hepatitis B infection and immunity is not exclusionary. Positive hepatitis C antibody with negative viral load or documented antiviral hepatitis C treatment with one post treatment non-detectable hepatitis C viral load is not exclusionary
* Recent significant blood or plasma donation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Transgender Female
Enrollment: 8 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Clinical Research Unit at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Pharmacokinetic data will be updated in study outcome and results.

REFERENCES:
- [Result] Lam K, Kraft WK, Zhan T, Lam E. Bidirectional pharmacokinetics of doravirine, tenofovir, and feminizing hormones in transgender women (IDentify): A randomized crossover trial. Clin Transl Sci. 2024 Mar;17(3):e13721. doi: 10.1111/cts.13721. PMID 38421210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through social media outreach and by interaction with advocacy groups. They were enrolled in the study between January 4, 2022 and September 21, 2022 at the Clinical Research Unit at Thomas Jefferson University.
Pre-assignment Details: 8 enrolled participants were randomized 1:1 to either Sequence E of F.
Groups:
- Sequence E: 4 of 8 enrolled participants were assigned to receive Sequence E, which consisted of Treatment A, B, and C administered during period I, II, and III, respectively.
  Treatment A: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate alone Treatment B: Single-dose estradiol and spironolactone co-administered with placebo Treatment C: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone Doravirine/Lamivudine/Tenofovir: 100mg/300mg/300mg orally for one dose, daily Spironolactone 100mg: 200mg orally for two doses, twice-daily Estradiol 2mg: 4mg orally for two doses, twice-daily Placebo: Placebo for one dose, daily
- Sequence F: 4 of 8 enrolled participants were assigned to receive Sequence F, which consisted of Treatment C, B, and A administered during period I, II, and III, respectively.
  Treatment A: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate alone Treatment B: Single-dose estradiol and spironolactone co-administered with placebo Treatment C: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone Doravirine/Lamivudine/Tenofovir: 100mg/300mg/300mg orally for one dose, daily Spironolactone 100mg: 200mg orally for two doses, twice-daily Estradiol 2mg: 4mg orally for two doses, twice-daily Placebo: Placebo for one dose, daily
Period: Overall Study
Arm/Group | Sequence E | Sequence F
Started | 4 | 4
Completed | 3 | 3
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: 8 participants were enrolled in the study and randomized 1:1 to either Sequence E or F.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence E | Sequence F | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 25.5 [25 to 38] | 27 [24 to 31] | 25.5 [24 to 38]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Transgender female (male-to-female) | 4 | 4 | 8
  Gender Identity: Transgender male (female-to-male) | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Doravirine Area Under the Plasma Concentration Versus Time Curve From 0 Hours to Infinity (AUC0-∞)
Description: Doravirine AUC derived from plasma sampling with geometric mean ratio compared between treatment arms
Time Frame: Pre-dose, 0.5, 1, 2, 6, 12, 24, 48, 72, 96 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Treatment C: Treatment C: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone
  Doravirine/Lamivudine/Tenofovir: 100mg/300mg/300mg orally for one dose, daily Spironolactone 100mg: 200mg orally for two doses, twice-daily Estradiol 2mg: 4mg orally for two doses, twice-daily
- Treatment A: Treatment A: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate alone
  Doravirine/Lamivudine/Tenofovir: 100mg/300mg/300mg orally for one dose, daily
Arm/Group | Treatment C | Treatment A
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 17798.14 (21.7) | 18413.21 (41.75)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratio for doravirine AUC falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; A post hoc power analysis determined 80% power would be achieved for 6 subjects to detect an effect size of 1.43 or greater at 5% significance level; Geometric mean ratio = 0.97, 90% CI 2-sided [0.76 to 1.24] — Ratio represents Treatment C (Single-dose oral doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone) over Treatment A (Single-dose oral doravirine/lamivudine/tenofovir disoproxil fumarate alone)

2. Primary Outcome: Doravirine Maximum Concentration (Cmax)
Description: Doravirine maximum observed concentration during the dosing interval with geometric mean ratio compared between treatment arms
Time Frame: Pre-dose, 0.5, 1, 2, 6, 12, 24, 48, 72, 96 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C | Treatment A
Number analyzed (Participants) | 6 | 6
ng/mL | 745.46 (21.43) | 799.67 (26.01)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratio for doravirine Cmax falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.93, 90% CI 2-sided [0.66 to 1.32] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Doravirine Trough Concentration (C24)
Description: Doravirine observed trough concentration during the dosing interval with geometric mean ratio compared between treatment arms
Time Frame: 24 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C | Treatment A
Number analyzed (Participants) | 6 | 6
ng/mL | 283.74 (25.42) | 292.89 (49.3)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratio for doravirine C24 falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.97, 90% CI 2-sided [0.76 to 1.24] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Tenofovir Disoproxil Fumarate Area Under the Plasma Concentration Versus Time Curve From 0 Hours to Infinity (AUC0-∞)
Description: Tenofovir AUC derived from plasma sampling with geometric mean ratio compared between treatment arms
Time Frame: Pre-dose, 0.5, 1, 2, 6, 12, 24, 48, 72, 96 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Treatment C | Treatment A
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 2370.6 (23.42) | 2031.84 (35.25)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratio for tenofovir AUC falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.17, 90% CI 2-sided [0.91 to 1.50] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Tenofovir Disoproxil Fumarate Maximum Concentration (Cmax)
Description: Tenofovir maximum observed concentration during the dosing interval
Time Frame: Pre-dose, 0.5, 1, 2, 6, 12, 24, 48, 72, 96 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C | Treatment A
Number analyzed (Participants) | 6 | 6
ng/mL | 178.84 (58.4) | 129.95 (99.92)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratio for tenofovir Cmax falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.38, 90% CI 2-sided [0.73 to 2.60] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Tenofovir Disoproxil Fumarate Trough Concentration (C24)
Description: Tenofovir observed trough concentration during the dosing interval with geometric mean ratio compared between treatment arms
Time Frame: 24 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment C | Treatment A
Number analyzed (Participants) | 6 | 6
ng/mL | 29.59 (24.23) | 26 (35.77)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratio for tenofovir C24 falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.14, 90% CI 2-sided [0.93 to 1.40] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Estradiol Area Under the Plasma Concentration Versus Time Curve From 0 Hours to Infinity (AUC0-∞)
Description: Estradiol area under the plasma concentration versus time curve from 0 hours to infinity (AUC) derived from plasma sampling
Time Frame: Pre-dose, 0.5, 2, 6, 12, 24, 48, 72, 96 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Groups:
- Treatment B: Treatment B: Single-dose estradiol and spironolactone co-administered with placebo
  Spironolactone 100mg: 200mg orally for two doses, twice-daily Estradiol 2mg: 4mg orally for two doses, twice-daily Placebo: Placebo for one dose, daily
Arm/Group | Treatment C | Treatment B
Number analyzed (Participants) | 6 | 6
hr*pg/mL | 9370.25 (14.36) | 9677.31 (43.29)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratio for estradiol AUC falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 0.97, 90% CI 2-sided [0.70 to 1.35] — Ratio represents Treatment C (Single-dose oral doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone) over Treatment B (Single-dose estradiol and spironolactone co-administered with placebo)

8. Primary Outcome: Estradiol Maximum Concentration (Cmax)
Description: Estradiol maximum observed concentration during the dosing interval with geometric mean ratio compared between treatment arms
Time Frame: Pre-dose, 0.5, 2, 6, 12, 24, 48, 72, 96 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment C | Treatment B
Number analyzed (Participants) | 6 | 6
pg/mL | 118.08 (20.5) | 105.14 (21.26)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratios for estradiol Cmax falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.12, 90% CI 2-sided [0.92 to 1.36] — [estimate comment as in outcome 7, analysis 1]

9. Primary Outcome: Estradiol Trough Concentration (C12)
Description: Estradiol observed trough concentration during the dosing interval with geometric mean ratio compared between treatment arms
Time Frame: 12 hours post-dose for all participants
Population: 6 participants completed the study and were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Treatment C | Treatment B
Number analyzed (Participants) | 6 | 6
pg/mL | 100.26 (26.56) | 92.01 (36.94)
Statistical Analysis 1: Comparison: Treatment C; 6 participants completed the study and were included in the pharmacokinetic analysis. As all participants received the same treatment groups but not necessarily in the same order, calculations were done between arms (Sequence E and F). 10 subjects was determined to achieve 80% power to reject the null hypothesis (geometric mean ratios for estradiol C12 falls outside of the no-effect boundaries) with two-sided significance level of 0.05 assuming a mean ratio of 1 for no effect; Test type: Equivalence — The no-effect (bioequivalence) boundaries of 80%-125% were used; A two-sided significance level of 0.05 with a mean ratio of 1 for no effect was assumed; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.09, 90% CI 2-sided [0.88 to 1.35] — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: 9 weeks, up to 30 days after last dose of drug administered
Description: Adverse events were collected throughout the duration of the study, up to 30 days after last dose of drug administered. All subjects received all treatments, and as such the comparisons are between sequences. Adverse events were not separated out by treatment, but only by Sequence. Adverse Events were monitored without regard to the specific intervention or period.
Groups:
- Sequence E: All subjects received all treatments, and as such the comparisons are between sequences.
  Adverse events were not separated out by treatment, but only by Sequence
  4 of 8 enrolled participants were assigned to receive Sequence E, which consisted of Treatment A, B, and C administered during period I, II, and III, respectively.
  Treatment A: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate alone Treatment B: Single-dose estradiol and spironolactone co-administered with placebo Treatment C: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone Doravirine/Lamivudine/Tenofovir: 100mg/300mg/300mg orally for one dose, daily Spironolactone 100mg: 200mg orally for two doses, twice-daily Estradiol 2mg: 4mg orally for two doses, twice-daily Placebo: Placebo for one dose, daily
- Sequence F: All subjects received all treatments, and as such the comparisons are between sequences.
  Adverse events were not separated out by treatment, but only by Sequence
  4 of 8 enrolled participants were assigned to receive Sequence F, which consisted of Treatment C, B, and A administered during period I, II, and III, respectively.
  Treatment A: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate alone Treatment B: Single-dose estradiol and spironolactone co-administered with placebo Treatment C: Single-dose oral Doravirine/lamivudine/tenofovir disoproxil fumarate co-administered with estradiol and spironolactone Doravirine/Lamivudine/Tenofovir: 100mg/300mg/300mg orally for one dose, daily Spironolactone 100mg: 200mg orally for two doses, twice-daily Estradiol 2mg: 4mg orally for two doses, twice-daily Placebo: Placebo for one dose, daily
Arm/Group | Sequence E | Sequence F
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sequence E (N=4) | Sequence F (N=4)
Nausea/vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Application site erythema (General disorders) | 0 | 1 — Tegaderm redness
Catheter site redness (General disorders) | 0 | 1
Catheter site pruritus (General disorders) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 — Muscle cramps
Brain fog (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Distractibility (Psychiatric disorders) | 1 | 0
Dysphoria (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1
Gender dysphoria (Psychiatric disorders) | 1 | 0
Libido increased (Psychiatric disorders) | 1 | 1
Mood swings (Psychiatric disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 1
Seborrhoea (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04283656/Prot_SAP_000.pdf